CLINICAL TRIAL: NCT00115700
Title: A Randomised Multicentre Trial of Involved Field Radiotherapy Versus Involved Field Radiotherapy Plus Chemotherapy in Combination With Rituximab (Mabthera®) for Stage I - II Low Grade Follicular Lymphoma
Brief Title: Radiotherapy Versus Radiotherapy Plus Chemotherapy in Early Stage Follicular Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Australasian Leukaemia and Lymphoma Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 99.03; ALLG NHLLOW5 (Other: Collaborative group)
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Follicular Lymphoma
Keywords: Radiotherapy; Chemotherapy; Rituximab; Randomised Trial; Stage I-II low grade follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Cyclophosphamide; Radiotherapy; Radiation; Vincristine; Prednisolone; Prednisone; Methylprednisolone; Rituximab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiotherapy+ Chemotherapy (Experimental): Involved field Radiotherapy (RT) 30-36 GY plus Cyclophosphamide, Vincristine and Prednisolone (CVP) + rituximab × 6 cycles
  Interventions: Drug: Cyclophosphamide; Radiation: Radiotherapy; Drug: Vincristine; Drug: Prednisolone; Drug: Rituximab
- Radiotherapy alone (Active Comparator): Involved field Radiotherapy (30-36 GY) alone
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cyclophosphamide — 1000 mg/m2 I.V. on day 1
  Other Names: Cycloblastin, Endoxan
  Arms: Radiotherapy+ Chemotherapy
Radiation: Radiotherapy — The prescribed dose to the target volume will be 30 Gy. Daily fractions of 1.5-2.0 Gy will be employed.
  Other Names: Radiation
Drug: Vincristine — 1.4 mg/m2 (maximum single dose of 2 mg) I.V. on day 1
  Other Names: Vincristine Sulfate Injection
  Arms: Radiotherapy+ Chemotherapy
Drug: Prednisolone — 50 mg/m2 orally daily for days 1 - 5
  Other Names: Panafcort, Panafcortelone, Predsone, Predsolone
  Arms: Radiotherapy+ Chemotherapy
Drug: Rituximab — 375 mg/m2 IV Infusion day 1
  Other Names: Erbitux, Mabthera
  Arms: Radiotherapy+ Chemotherapy

SUMMARY:
Patients with stage I and II low grade follicular lymphoma are randomised between standard therapy (involved field radiotherapy) and investigational therapy (involved field radiotherapy and chemotherapy plus rituximab). The main endpoint is progression free survival but overall survival and the influence of t(14;18) status will also be studied.

DETAILED DESCRIPTION:
Radiotherapy is the only modality which has been proven to have curative potential in patients with localised low grade lymphoma. Despite excellent control of the local tumour, most patients relapse outside the area treated with radiation and most of these ultimately die from lymphoma. This study tests the hypothesis that the addition of six cycles of chemotherapy plus rituximab (systemic chemotherapy) can eradicate undetectable lymphoma deposits outside the radiation field and thereby improve the cure rate. The study will specifically test the hypothesis that six cycles of adjuvant CVP chemotherapy (cyclophosphamide, vincristine, prednisolone) in combination with Rituximab will improve progression-free survival for patients with stage I and II low-grade follicular lymphoma treated with involved-field radiotherapy (IFRT). That is, will patients given radiotherapy plus systemic chemotherapy live longer or remain free from disease longer than patients treated with radiation alone? Radiotherapy alone is widely regarded as the standard treatment for this disease.

There are a number of secondary endpoints to the study, as follows:

1. Comparison the pre- and post-treatment prevalence of the t(14:18) translocation, in peripheral blood and bone marrow, of patients treated with either IFRT alone or IFRT plus chemotherapy. This translocation is potentially a marker for minimal residual disease and eradication of the marker from blood cells may have prognostic implications. The clinical value of "molecular remission" as an early predictor of freedom from progression (FFP) and survival will be assessed.
2. Comparison of overall survival and FFP for patients treated with IFRT alone with overall survival and FFP for patients treated with combined IFRT and systemic therapy. Delay of progression of disease may be of limited value if overall survival is the same.
3. Comparison of acute and late toxicity and second malignancy rates for patients treated with IFRT or IFRT plus systemic therapy.
4. Delineation of the location of first relapse in relation to radiation therapy fields.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) with histologically documented "follicular lymphoma, grade 1", grade 2", or "follicular lymphoma, grade 3a" diagnosed following an excisional, incisional or generous core biopsy. (i.e. an FNA alone is insufficient.)
* Disease limited to stages I and II after adequate staging
* Anticipated life expectancy > 5 years
* Given written informed consent
* Been assessed by a radiation oncologist and a medical oncologist/ haematologist
* WCC > 3.0 x 10^9/L, platelet count > 100 x 10^9/L, serum creatinine < 0.15 mmol/L
* Ability to commence radiotherapy within 6 weeks of randomisation
* Women using effective contraception, are not pregnant and agree not to become pregnant during participating in the trial and during the 12 months thereafter. Men agree not to father a child during participation in the trial and during the 12 months thereafter.

Exclusion Criteria:

* Received previous systemic cytotoxic chemotherapy.
* Received previous radiotherapy, (except superficial radiation therapy for non-melanoma skin cancers).
* Received previous immunotherapy.
* A medical contraindication to radiotherapy, chemotherapy, or rituximab.
* Any previous or concurrent malignancy other than curatively treated non-melanoma skin cancer, level 1 malignant melanoma, or in situ cervical cancer, unless disease and treatment-free for 5 years.
* Such extensive involvement of the thorax that treatment with radiation therapy alone would be hazardous because of excessive lung irradiation, even if a shrinking field technique were employed.
* Suspected or confirmed pregnancy. Must not be lactating.
* Patients who have known human immuno-deficiency virus (HIV) infection or active hepatitis B (HBV).
* Treatment within a clinical study within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2000-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS). Period from the date of randomisation to 1st progression of disease or death from any cause. | Main analysis after at least 3 years of follow-up following the end of accrual. An updated analysis may be done on completion of 5 years follow-up after the end of accrual. Long term follow-up analysis is planned after 10 years of follow-up

SECONDARY OUTCOMES:
Pre- and post-treatment prevalence of the t(14;18) translocation, in peripheral blood and bone marrow between arms | Peripheral blood at commencement of treatment, after 1 year and upon relapse is collected and stored for later analysis to be done as part of translational studies when funding becomes available
Overall Survival (OS) | Main analysis will be done on completion of 5 years follow-up after the end of accrual. An interim analysis to be done after at least 3 years of follow-up. A futility analysis will be performed after the 5 year analysis. In the absence of futility being
  Period from date of randomisation to date of death from any cause.
Location of first relapse | Main analysis after at least 3 years of follow-up following the end of accrual. An updated analysis may be done on completion of 5 years follow-up after the end of accrual
  Period from date of randomisation to date of first relapse location via CT scan and or other imaging as required
To compare time to evolution to higher histological grade | Main analysis after at least 3 years of follow-up following the end of accrual. An updated analysis may be done on completion of 5 years follow-up after the end of accrual
  Period from date of randomisation to date of higher histological grade via CT scan and or other imaging as required
Freedom from progression. | Main analysis after at least 3 years of follow-up following the end of accrual. An updated analysis may be done on completion of 5 years follow-up after the end of accrual. Long term follow-up analysis is planned after 10 years of follow-up
  Period from date of randomisation to date of first disease progression.
Acute and late toxicities and secondary malignances | Frame after at least 3 years of follow-up following the end of accrual. An updated analysis may be done on completion of 5 years follow-up after the end of accrual

CONTACTS AND LOCATIONS:
Overall Officials: Michael MacManus, MD, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (21):
- Australia (17):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Albury Base/Murray Valley Private Hospital, West Albury, New South Wales
  - Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Radiation Oncology - Mater Centre, South Brisbane, Queensland
  - Genesis Cancer Care (previously Premion), Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - St John of God Hospital, Ballarat, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Princess Margaret Hospital, Toronto, Canada
- New Zealand (3):
  - Auckland Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington

REFERENCES:
- [Derived] MacManus M, Fisher R, Roos D, O'Brien P, Macann A, Davis S, Tsang R, Christie D, McClure B, Joseph D, Jayamohan J, Seymour JF. Randomized Trial of Systemic Therapy After Involved-Field Radiotherapy in Patients With Early-Stage Follicular Lymphoma: TROG 99.03. J Clin Oncol. 2018 Oct 10;36(29):2918-2925. doi: 10.1200/JCO.2018.77.9892. Epub 2018 Jul 5. PMID 29975623
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au